CLINICAL TRIAL: NCT06510478
Title: Efficacy of Group Life Skill Intervention to Enhance Well-Being Among Higher Education Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Kiran Mushtaq, Efficacy of Group Life Skill Intervention to enhance Well-Being among Higher Education Students, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FJWU/EC/2023/66
Record Dates: First submitted 2024-07-13; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Psychological Distress; Mental Health Issue; Quality of Life; Well-Being, Psychological
Keywords: Efficacy; Group Life Skill Intervention; Psychological Distress; Life skills; Quality of Life; Well being
MeSH Terms: conditions — Psychological Well-Being | interventions — Therapeutics; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): Who receives intervention. Life Skill intervention will be administered in 12 sessions.
  Interventions: Behavioral: Group Life Skill Intervention
- Control Group (Placebo Comparator): Who do not receive any intervention.
  Interventions: Behavioral: Treatment as Usual for Control Group
- Waitlist Control Group (Active Comparator): Who are on the waitlist and will receive intervention components if the intervention is proven to be effective.
  Interventions: Behavioral: Group Life Skill Intervention

INTERVENTIONS:
Behavioral: Group Life Skill Intervention — This 13-session life skills program covers essential topics in one-hour sessions. It starts with introductions and team building, then progresses through leadership, self-esteem, communication, stress management, positive thinking, confidence building, volunteering, decision-making, problem-solving, conflict resolution, and negotiation. Each session includes ice-breakers, discussions, and targeted exercises. Each session incorporates ice-breakers, open discussions, and targeted exercises to ensure active learning and skill internalization. Duration of each session was 1 hour.
  Arms: Intervention Group; Waitlist Control Group
Behavioral: Treatment as Usual for Control Group — Standard psychological interventions i.e. Debreathing, Meditation, supportive counseling, or psychoeducation.
  Arms: Control Group

SUMMARY:
The primary aim of this study is to investigate the Efficacy of Group life skills intervention designed to improve the well-being, Life skills, and Quality of life of higher education students. The study also identifies the feasibility of the Life skill intervention in the context of Pakistan. We will also compare these outcomes between two groups: one receiving the intervention and the other not receiving any treatment.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the Efficacy of Group life skills intervention designed to improve the well-being, Life skills, and Quality of life of higher education students. The study also identifies the feasibility of the Life skill intervention in the context of Pakistan. We will also compare these outcomes between two groups: one receiving the intervention and the other not receiving any treatment.

Study Tasks:

Participants, who are University Students aged 21-30 years, were asked to provide informed consent to participate in the study. They completed questionnaires to assess their Life skills, Psychological distress, Well-being, and Quality of life as a pre-assessment.

Participants in the intervention group undergo the Life Skill Intervention, which includes activities like Team building skills, Leadership Skills, Self-respect and appreciation, Effective Communication Skills, Dealing with stress, Positive Thinking, Enhancing confidence, Volunteering, Decision Taking, Problem Solving, Conflict Resolution, Negotiating.

After the intervention, participants completed a post-assessment questionnaires to measure changes in Life skills, Psychological distress, Well-being, and Quality of life.

There will be a control group that does not receive any treatment.

Comparison Group:

Researchers compared the outcomes between the intervention group, who received the Life Skill Intervention and the control group, who did not receive any treatment. This will help us determine if the intervention had a significant impact on Life skills, Psychological distress, Well-being, and Quality of life outcomes for University students.

ELIGIBILITY:
Inclusion Criteria:

* Students of public sector university of Pakistan.
* Students aged 21-30.
* Students accessed with decreased psychological well-being.

Exclusion Criteria:

* Students of private universities in Pakistan
* Students with any physical disability.
* Students having a prior history of psychiatric illness.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Well Being | 2 Months
  14-item scale 'Warwick-Edinburgh Mental Well-being Scale' used to measure. Minimum score on this scale is 0 and maximum score is 30.Higher score would indicate higher level of well being.

SECONDARY OUTCOMES:
Life Skills | 2 Months
  14-item scale- Life skills questionnaire used to measure. The minimum score on this scale is 14 and the maximum score is 70. Scoring higher on this scale indicates higher life skills in individuals.
Psychological Distress | 2 Months
  Depression, Anxiety, and Stress Scale used to measure. The minimum score on this scale is 0 and the maximum score is 63. Higher scores on all subscales indicate a higher level of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Mushtaq, PhD Scholar, Principal Investigator — Fatima Jinnah Women University
Locations (1):
- University of Sahiwal, Sahiwal, Punjab Province, Pakistan